CLINICAL TRIAL: NCT03533088
Title: Comparing Two Different Rehabilitation Protochols on Patients With Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Irem Duzgun, Doç. Dr. İrem Düzgün, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1233412334
Record Dates: First submitted 2018-05-10; First posted 2018-05-22 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Rotator Cuff Tear
Keywords: shoulder; rotator cuff; exercise
MeSH Terms: conditions — Rotator Cuff Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospitalized rehabilitation (Experimental): Patients in this group will recieve rehabilitation program twice in a week at our clinic after the surgical procedure until post-operative 12 weeks.
  Interventions: Other: Hospitalized rehabilitation
- Home-based rehabilitation (Experimental): Patients in his groups will performed home-based rehabilitation in the early stages of the post-op period. They will com to our clinic once in a two weeks and the recieve the exercise program to perform at home until the 6. weeks of the post-operative period. After the 6. week they will come to our clinic once in a week until the post-operative 12. week.
  Interventions: Other: Home-based rehabilitation

INTERVENTIONS:
Other: Hospitalized rehabilitation — Patients will recive a rehabilitation prgram at the clinic twice in a week until the post-operative 12. weeks
  Arms: Hospitalized rehabilitation
Other: Home-based rehabilitation — Patients will recive a home program once in a two weeks until the 6. weeks of post-operative period. Then will start to recieve a rehabilitation program ar the clinic once in a week auntil the 12. week of the post-operative period.
  Arms: Home-based rehabilitation

SUMMARY:
Rotator cuff (RC) repair is one of the most common treatment approch to relief the pain and improve the shoulder function on patients with rotator cuff rupture. Despite the improved surgical techniques and decreased failure rate, there are still complications after the surgey like shoulder persistant shoulder pain, stiffness even re-tear. Therefore, rehabilitation after the RC repair procedure is crucial for the success of the treatment. However, there is no concencus between the post-operative rehabilitation protochol. The aim of this study is to compare two different rehabilitation protochols on patients with RC repair.

DETAILED DESCRIPTION:
Rotator cuff (RC) repair is one of the most common treatment approch to relief the pain and improve the shoulder function on patients with rotator cuff rupture. Despite the improved surgical techniques and decreased failure rate, there are still complications after the surgey like shoulder persistant shoulder pain, stiffness even re-tear. Therefore, rehabilitation after the RC repair procedure is crucial for the success of the treatment. However, there is no concencus between the post-operative rehabilitation protochol. The aim of this study is to compare two different rehabilitation protochols in terms of shoulder range of motion, self-reported shoulder function and pain on patients with RC repair.

ELIGIBILITY:
Inclusion Criteria:

* Having a Rotator Cuff repair surgery
* Having post-op rehabilitation program at our clinic until post-op 3 months
* No previous surgery in the shoulder joint

Exclusion Criteria:

* Additional pathology other then RC tear
* Refusing to participate to the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
scapular kinematics | 6 months
  3-Dimensional scapular kinematics will be assessed

SECONDARY OUTCOMES:
gleno-humeral range of motion | 6 months
  patients' shoulder range of motions will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Taha Yıdız, Msc, Study Chair — İnvestigator
Locations (1):
- Hacettepe Univercity, Faculty of Physical Theraphy and Rehablitation, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gallagher BP, Bishop ME, Tjoumakaris FP, Freedman KB. Early versus delayed rehabilitation following arthroscopic rotator cuff repair: A systematic review. Phys Sportsmed. 2015 May;43(2):178-87. doi: 10.1080/00913847.2015.1025683. Epub 2015 Mar 22. PMID 25797067
- [Result] Thomson S, Jukes C, Lewis J. Rehabilitation following surgical repair of the rotator cuff: a systematic review. Physiotherapy. 2016 Mar;102(1):20-8. doi: 10.1016/j.physio.2015.08.003. Epub 2015 Sep 8. PMID 26510584